CLINICAL TRIAL: NCT03559049
Title: A Phase I/II Multi-site Study of Rucaparib and Pembrolizumab Maintenance Therapy in Stage IV Non-Squamous Non-Small Cell Lung Cancer After Initial Therapy With Carboplatin, Pemetrexed, and Pembrolizumab
Brief Title: Rucaparib and Pembrolizumab for Maintenance Therapy in Stage IV Non-Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to financial hardships suffered by the stakeholder
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.033; HUM00142973 (Other: University of Michigan)
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib and Pembrolizumab Maintenance (Experimental): All patients will receive induction therapy with Pembrolizumab (200mg IV on day 1 of every 21 days), Pemetrexed (500mg/m^2 IV on day 1 of every 21 days), and Carboplatin (AUC5 IV on day 1 of every 21 days).
  This will be followed by maintenance therapy with Pembrolizumab (200mg IV on day 1 of every 21 days) and Rucaparib (600mg PO BID days 1-21 of each 21 day cycle).
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Rucaparib

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV every 21 days
Drug: Pemetrexed — 500mg/m^2 IV every 21 days
Drug: Carboplatin — AUC 5 IV every 21 days
Drug: Rucaparib — 600mg PO, BID days 1-21 of each 21 day cycle

SUMMARY:
This study is a multi-center, Phase I/II, single arm trial to assess the safety and efficacy of the combination of oral rucaparib plus intravenous pembrolizumab as maintenance therapy in patients with stage IV non-squamous non-small cell lung cancer (NSCLC) without progressive disease (PD), as confirmed on CT scans, after induction therapy with carboplatin/pemetrexed/pembrolizumab (CPP) triplet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Have a life expectancy of at least 3 months.
* Have a diagnosis of stage IV non-squamous NSCLC whose tumors do not have an epidermal sensitizing growth factor (EGFR) mutation or BRAF mutation or rearrangements in ALK (anaplastic lymphoma kinase) or ROS-1 and have at least one measurable lesion based on RECIST v1.1.
* Have a performance status of 0 or 1 on the ECOG Performance Scale (Appendix 15.1).
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a serum pregnancy test within -28 days of enrollment and 72 hours prior to receiving the first dose of study medications.
* Female subjects of childbearing potential must be willing to use a highly effective method of contraception as outlined in Section 6.3.3 for the course of the study through 180 days after the last dose of study medications. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 6.3.3, starting with the first dose of study therapy through 180 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* If the patient has archival tissue, this should be collected for correlative studies. If archival tissue does not exist, a new biopsy is not required

Exclusion Criteria:

* Received previous systemic therapy for stage IV NSCLC
* Received radiation to the lungs >30Gy ≤6 months of enrollment
* Received palliative radiation within 7 days of enrollment
* Had prior treatment with any other anti-PD-1, PD-L1, or PD-L2 agent or an antibody targeting other immune-regulatory receptors or mechanisms
* Received prior treatment with a PARP inhibitor
* Has a known history of prior malignancy except if the patient has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment within the past 2 years
* Subjects requiring daily corticosteroids >10mg of prednisone (or its equivalent) would be excluded from the study.
* Has evidence of interstitial lung disease or a history of non-infectious pneumonitis that required oral or intravenous glucocorticoids to assist with management
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with informed consent through 180 days after the last dose of trial treatment
* Has a diagnosis of immunodeficiency (including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency (AIDS)-related illness) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment
* Has a known history of active TB (Bacillus Tuberculosis)
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of enrollment
* A medical condition that requires daily systemic corticosteroids, greater than the equivalent of 10mg of prednisone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Qin, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - The University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was deemed an incorrect consent after enrollment and never started on therapy
Groups:
- Rucaparib and Pembrolizumab Maintenance: All patients received induction therapy with Pembrolizumab (200mg IV on day 1 of every 21 days), Pemetrexed (500mg/m^2 IV on day 1 of every 21 days), and Carboplatin (AUC5 IV on day 1 of every 21 days).
  This was followed by maintenance therapy with Pembrolizumab (200mg IV on day 1 of every 21 days) and Rucaparib (600mg PO BID days 1-21 of each 21 day cycle).
  Pembrolizumab: 200mg IV every 21 days
  Pemetrexed: 500mg/m^2 IV every 21 days
  Carboplatin: AUC 5 IV every 21 days
  Rucaparib: 600mg PO, BID days 1-21 of each 21 day cycle
Period: Overall Study
Arm/Group | Rucaparib and Pembrolizumab Maintenance
Started | 24
Completed | 10
Not Completed | 14
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — Sponsor termination | 3

BASELINE CHARACTERISTICS:
Population: 1 patient was deemed an incorrect consent after enrollment and never started on therapy
Arm/Group | Rucaparib and Pembrolizumab Maintenance
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Median Duration of Time From Start of Treatment to Time of Progression
Description: The primary endpoint is median progression free survival (PFS) which is defined as the median duration of time from the start of treatment to progression. Progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Up to 5 years
Population: Per the protocol, the Evaluable population is those patients who received at least one cycle of maintenance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Pembrolizumab Maintenance
Number analyzed (Participants) | 14
months | 10.6 [8.3 to NA] — The upper confidence limit for the median could not be estimated because there were too few progression events. The upper confidence limit curve never reaches 50 percent, so the upper confidence limit is not estimable.

2. Secondary Outcome: Median Duration of Time From the Start of Treatment Until Death
Description: The secondary endpoint is median overall survival (OS) which is defined as the median duration of time from the start of treatment until death.
Time Frame: Up to 5 years
Population: Per the protocol, the Evaluable population is those patients who received at least one cycle of maintenance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Pembrolizumab Maintenance
Number analyzed (Participants) | 14
months | 37.6 [25.6 to NA] — The upper confidence limit for the median could not be estimated because there were too few progression events. The upper confidence limit curve never reaches 50 percent, so the upper confidence limit is not estimable.

3. Secondary Outcome: Response Rate
Description: Percentage of patients who achieve a complete or partial response after at least one cycle of maintenance therapy with rucaparib and pembrolizumab. Response assessed by immune-related Response Evaluation Criteria in Solid Tumors (irRecist).
Time Frame: Up to 5 years
Population: Per the protocol, the Evaluable population is those patients who received at least one cycle of maintenance.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib and Pembrolizumab Maintenance
Number analyzed (Participants) | 14
Participants | 9

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days (non-serious) and 90 days (serious) after the last dose of study treatment. Data was collected up to 5 years.
Description: Per the protocol, the Evaluable population is those patients who received at least one cycle of maintenance.
Arm/Group | Rucaparib and Pembrolizumab Maintenance
All-Cause Mortality (participants affected / at risk) | 7/14
Serious Adverse Events (participants affected / at risk) | 8/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib and Pembrolizumab Maintenance (N=14)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Fall (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Urosepsis
Lung infection (Infections and infestations) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib and Pembrolizumab Maintenance (N=14)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Flank pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — decreased appetite
Nausea (Gastrointestinal disorders) | 3 (6)
Pain (General disorders) | 2 (4)
Pain in extremity (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Dysuria
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Covid-19
Sinusitis (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (2)
Weight gain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating Site agrees not to publish or publically present the Study Data or Study Results, until Michigan or Michigan's Investigator has first Published the Study Data or Study Results. Thereafter, Participating Site may publish or publically present the Study Data and/or Study Results. If Michigan has not Published the Study Data or Study Results within 12 months after the abandonment or termination of the Study, Participating Site may publish or present the Study Data or Study Results

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03559049/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03559049/ICF_001.pdf